CLINICAL TRIAL: NCT03778671
Title: Dexmedetomidine Versus Fentanyl Added to Levobupivacaine for Transversus Abdominis Plane (TAP) Block in Elderly Patients Undergoing Lower Abdominal Surgery
Brief Title: Dexmedetomidine Versus Fentanyl Added to Levobupivacaine for Transversus Abdominis Plane (TAP) Block
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17300222
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Transversus Abdominis Block
Keywords: transversus abdominis plane block; Dexmedetomidine; Fentanyl
MeSH Terms: interventions — Levobupivacaine; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group B (Experimental): Patients will receive Levobupivacaine 5%
  Interventions: Drug: Levobupivacaine
- Group D (Active Comparator): Patients will receive Levobupivacaine 5% + 1 µg/kg dexmedetomedine .
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Group F (Active Comparator): Patients will receive Levobupivacaine 5% + 1µg/kg fentanyl
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: Levobupivacaine — Patients will receive Levobupivacaine 5%
  Other Names: Levobupivacaine hydrate
  Arms: Group B
Drug: Dexmedetomidine Injection [Precedex] — Patients will receive Levobupivacaine 5% + 1 µg/kg dexmedetomedine
  Arms: Group D
Drug: fentanyl — Patients will receive Levobupivacaine 5% + 1 µg/kg fentanyl
  Arms: Group F

SUMMARY:
The perioperative management of pain following lower abdominal surgery can pose a challenge to anesthesia providers. Conventional practice has involved the use of opioids as well as neuraxial analgesic techniques. Unfortunately, these therapies are not without potential risks and side effects. These include nausea, vomiting, pruritus, urinary retention, constipation, respiratory depression, and sedation.

DETAILED DESCRIPTION:
One method used in this multimodal approach is the transversus abdominis plane block. This block, as first described by Rafi. in 2001, provides analgesia to the anterolateral abdominal wall. In 2007, McDonnell et al. further studied this technique in patients undergoing large-bowel resection. He discovered a reduction in postoperative pain and morphine consumption in the first 24 hours postoperatively, resulting in fewer opioid mediated side effects. In this same year, Hebbard et al. described the use of ultrasound guidance to provide real-time imaging of the muscle layers and needle placement to improve transversus abdominis plane block accuracy. In 2008, Hebbard. described the subcostal approach of transversus abdominis plane block, to target the nerves of the upper abdomen. Transversus abdominis plane blocks continue to be studied and developed as an effective method for providing analgesia for numerous types of transverses abdominis plane block duration is limited to effect of administered local anesthetics.The use of an infusion catheter to administer local anesthetics is an option to prolong the block's duration. Recently, adjuvant medications were added to local anesthetics to prolong the effect of transverses abdominis plane block .

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status II-III,
* scheduled for uncomplicated elective paraumbilical hernia repair.

Exclusion Criteria:

1. Patient refusal to participate in the study
2. Patients with coagulopathy or under anticoagulation therapy.
3. Infection near the site of needle insertion.
4. Body mass index > 40kg/m2
5. Patients with any neurological or neuromuscular disorder or history of seizures.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
first analgesic request | 24 hours
  first time to call for analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elvir-Lazo OL, White PF. The role of multimodal analgesia in pain management after ambulatory surgery. Curr Opin Anaesthesiol. 2010 Dec;23(6):697-703. doi: 10.1097/ACO.0b013e32833fad0a. PMID 20847690
- [Background] White PF, Kehlet H. Improving postoperative pain management: what are the unresolved issues? Anesthesiology. 2010 Jan;112(1):220-5. doi: 10.1097/ALN.0b013e3181c6316e. No abstract available. PMID 20010418
- [Background] Sharma P, Chand T, Saxena A, Bansal R, Mittal A, Shrivastava U. Evaluation of postoperative analgesic efficacy of transversus abdominis plane block after abdominal surgery: A comparative study. J Nat Sci Biol Med. 2013 Jan;4(1):177-80. doi: 10.4103/0976-9668.107286. PMID 23633858
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Aditianingsih D, Mochtar CA, Chandra S, Sukmono RB, Soamole IW. Comparison of Three-Quadrant Transversus Abdominis Plane Block and Continuous Epidural Block for Postoperative Analgesia After Transperitoneal Laparoscopic Nephrectomy. Anesth Pain Med. 2018 Sep 3;8(5):e80024. doi: 10.5812/aapm.80024. eCollection 2018 Oct. PMID 30533391